CLINICAL TRIAL: NCT04115735
Title: Obtaining His Bundle Recording From the Subclavian Vein in Patients Undergoing Permanent Pacemaker Implantation
Brief Title: His Bundle Recording From Subclavian Vein
Status: Terminated | Type: Observational
Why Stopped: Enrollment not feasible
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 18-109
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation; Congestive Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
His bundle pacing has been proposed as a superior alternative to standard right ventricular pacing. The purpose of this study is to investigate whether obtaining a His Bundle recording from the subclavian vein using a stylet driven pacemaker lead and commercially available sheath can be done in a quick and reliable manner. This would support the use of stylet driven leads for His bundle pacing.

DETAILED DESCRIPTION:
The purpose of this prospective observational study is to investigate whether obtaining a His Bundle recording from the subclavian vein using a stylet driven pacemaker lead and commercially available sheath can be done in a quick and reliable manner. Included in the study are patients undergoing permanent pacemaker implantation at Good Samaritan and Bethesda North Hospitals. The main outcome is successful recording of a His bundle potential. Secondary outcomes are the time necessary to record the His bundle and the measurement of the pacing threshold.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Male or Female Patients undergoing HIS bundle recording from the subclavian vein using a stylet driven pacemaker lead and commercially available sheath

Exclusion Criteria:

Patients who are unwilling or unable to sign the informed consent Pregnant women

Ages: 18 Years to 105 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing permanent pacemaker implantation identified by the TriHealth Heart Institute Electrophysiologists
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Successful recording of a His bundle potential | From beginning of procedure to the end
  The pacing lead will be connected to a standard EP recording system (GE CardioLab, LS Pro, or EP Med) a copy of the intracardiac electrograms demonstrating His bundle recording will be saved electronically.

SECONDARY OUTCOMES:
Time necessary to record the HIS bundle | From insertion of the pacing lead until successful measurement of HIS bundle
  Both the procedural and fluoroscopy time from insertion of the pacing lead until successful measurement of the His bundle
Pacing threshold | From beginning of procedure to the end of procedure
  Threshold will be measured in volts at 1 millisecond and recorded for selective His bundle capture, non-selective His bundle capture, and ventricular septal capture as appropriate for each patient. The measurement of a normal His Bundle threshold is < 2.0 V at 1.0 ms.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Winner, MD, Principal Investigator — TriHealth Heart Institute
Locations (1):
- TrIHealth, Cincinnati, Ohio, United States